CLINICAL TRIAL: NCT04302064
Title: A Randomized, Double-Blinded, Placebo-Controlled, Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-Ascending and Multiple Doses of ION-682884 in Healthy Japanese Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-Ascending and Multiple Doses of Eplontersen (Formerly Known as ION-682884, IONIS-TTR-LRx and AKCEA-TTR-LRx) in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ION-682884-CS20
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — eplontersen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplontersen (Experimental): Single dose on Day 1 or multiple doses (every 4 weeks for 12 weeks) of Eplontersen administered SC.
  Interventions: Drug: Eplontersen
- Placebo (Placebo Comparator): Single dose on Day 1 or multiple doses (every 4 weeks for 12 weeks) of Eplontersen-matching placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplontersen — Eplontersen administered SC
  Other Names: ION-682884; AKCEA-TTR-LRx; IONIS-TTR-LRx
  Arms: Eplontersen
Drug: Placebo — Eplontersen-matching placebo administered SC
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of single and potentially multiple doses of Eplontersen administered subcutaneously (SC) to healthy Japanese participants.

DETAILED DESCRIPTION:
This is a single-center, double-blinded, placebo-controlled study in up to 44 participants. Participants will be randomized to receive three subcutaneous single-ascending doses and potentially multiple doses of Eplontersen or placebo.

ELIGIBILITY:
Inclusion Criteria

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements
2. Healthy Japanese males or females of non-childbearing potential, aged 20 to 65 inclusive at the time of informed consent defined as being of first- or second-generation ethnic origin with each set of parents qualifying as Japanese under the prior generation. Generations will be defined as follows:

   * First generation Japanese participants must be born in Japan, cannot have lived outside of Japan for more than 10 years, must maintain Japanese diet, culture and lifestyle and parents and both sets of grandparents are of Japanese origin
   * Second-generation Japanese are participants who are born outside of Japan to the first-generation Japanese parents
3. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal (defined as 12 months of spontaneous amenorrhea without an alternative medical cause and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved Males must be surgically sterile or abstinent*, if engaged in sexual relations with a female of child-bearing potential, the participant must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 91 days (single-dose cohorts) or 13 weeks (multiple-dose cohorts) after the last dose of Study Drug (Eplontersen or placebo)

   * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception.
4. Willingness to take vitamin A supplements

Exclusion Criteria

1. Clinically significant abnormalities in medical history (e.g., previous acute coronary syndrome within 6 months of Screening, major surgery within 3 months of Screening) or physical examination
2. Screening laboratory results as follows, or any other clinically significant abnormalities in Screening laboratory values that would render a participant unsuitable for inclusion

   * Random spot urine protein/creatinine (P/C) ratio (UPCR) ≥ 200 milligrams per gram (mg/g).
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, alkaline phosphatase (ALP), serum creatinine, blood urea nitrogen (BUN) > upper limit of normal (ULN)
   * Fasting blood glucose > ULN
   * Platelet count < lower limit of normal (LLN)
3. Uncontrolled hypertension (blood pressure [BP] > 160/100 millimeters of mercury [mm Hg])
4. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at Least One Treatment-emergent Adverse Event (TEAE), Graded by Severity | Up to 92 days
Percentage of Participants with TEAEs Potentially Related to Study Drug | Up to 92 days
Percentage of Participants with Changes in Clinically Significant (CS) Laboratory Value Abnormalities | Up to 92 days

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diep JK, Yu RZ, Viney NJ, Schneider E, Guo S, Henry S, Monia B, Geary R, Wang Y. Population pharmacokinetic/pharmacodynamic modelling of eplontersen, an antisense oligonucleotide in development for transthyretin amyloidosis. Br J Clin Pharmacol. 2022 Dec;88(12):5389-5398. doi: 10.1111/bcp.15468. Epub 2022 Aug 7. PMID 35869634